CLINICAL TRIAL: NCT06567158
Title: The Impact of Carbohydrate Restriction on Glycemic Control in Children and Adolescents With Type 1 Diabetes Using a Hybrid Closed-loop Insulin Delivery System: a Randomized Cross-over Study
Brief Title: The Impact of a Moderate Carbohydrate Diet in Children With Type 1 Diabetes on Hybrid Closed-loop Therapy
Acronym: COMBINE1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: S68499
Record Dates: First submitted 2024-08-14; First posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: The study will be preceded by a screening period to check which participants are eligible for the study and a two-week run-in period during which, participants will be asked to document their eating patterns for one week in a digital food diary to base the moderate carbohydrate diet on.
  Participants will be randomized into two groups (1:1). One group will start at baseline with the traditional diet and after four weeks they will cross-over to the moderate carbohydrate diet for four weeks. The second group will start at baseline with the moderate carbohydrate diet and after four weeks they will crossover to the traditional diet for four weeks. Between the two diet periods there will be a wash-out period of six weeks.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: 1st Traditional diet, 2nd Moderate carbohydrate diet (Experimental): The group that starts with the traditional diet in the first 4-week diet period. After wash-out, this group will start with the moderate carbohydrate diet in the second 4-week diet period.
  Interventions: Other: Moderate carbohydrate diet; Other: Traditional diet
- Group 2: 1st Moderate carbohydrate diet, 2nd Traditional diet (Experimental): The group that starts with the traditional diet in the first 4-week diet period. After wash-out, this group will start with the moderate carbohydrate diet in the second 4-week diet period.
  Interventions: Other: Moderate carbohydrate diet; Other: Traditional diet

INTERVENTIONS:
Other: Moderate carbohydrate diet — During the moderate carbohydrate diet, participants will be asked to limit his/her carbohydrate intake to no more than 30% of their total energy intake.
Other: Traditional diet — During the traditional diet, participants do not follow any diet, however their carbohydrate intake must be at least 50% of their total energy intake.

SUMMARY:
In the past, carbohydrate restriction was indicated as a treatment for people with type 1 diabetes when exogenous insulin was not available. Now it is mainly used as an added treatment for people with type 1 diabetes on top of standard insulin administration and glucose monitoring. Despite previous studies, the impact of carbohydrate restriction on glycemic control and quality of life is still not clear. Furthermore, few studies exist on carbohydrate restriction in children with type 1 diabetes and combined with the use of hybrid closed-loop insulin delivery. Therefore this study will determine the impact on glycemic control and the feasability of a moderate carbohydrate diet compared to a traditional diet in children (7-17 years) with type 1 diabetes on top of using a hybrid closed-loop system. In this randomized, crossover study, 28 children will follow a moderate carbohydrate diet (four weeks) and a traditional diet (four weeks) in randomized order. With a run-in period (two weeks) prior to the first diet and a wash-out period (six weeks) between the two diets, the children will participate in the study for a total of 16 weeks. The primary endpoint is the difference of time spent in target range (defined as a sensor glucose value between 70 and 180 mg/dL) between the four-week moderate carbohydrate diet and the four-week traditional diet.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent (ICF) (both children/adolescents and parents)
* ≥7 and ≤17 years old at moment of ICF signature
* ≥6 months type 1 diabetes diagnosis at moment of ICF signature
* ≥3 months use of the hybrid closed-loop system Medtronic MiniMedTM 780G, Tandem t:slim X2 Control-IQTM or Mylife Ypsopump with CamAPS algorithm at moment of ICF signature
* Ability to understand, read, write and speak Dutch, French or English at moment of ICF signature

Exclusion Criteria:

* <7 or >17 years old at moment of ICF signature
* <6 months type 1 diabetes diagnosis at moment of ICF signature
* <3 months use of the advanced hybrid closed-loop system Medtronic MiniMedTM 780G, Tandem t:slim X2 Control-IQTM or Mylife Ypsopump with CamAPS algorithm at moment of ICF signature
* Any other insulin therapy than advanced hybrid closed-loop system Medtronic MiniMedTM 780G , Tandem t:slim X2 Control-IQTM or Mylife Ypsopump with CamAPS algorithm at moment of ICF signature
* Failure to understand, read, write or speak Dutch, French or English at moment of ICF signature

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Time in range | 4 weeks moderate carbohydrate diet and 4 weeks traditional diet
  Difference of time spent in range (70-180 mg/dL) between the moderate carbohydrate diet and the traditional diet.

SECONDARY OUTCOMES:
Time in tight range | 4 weeks moderate carbohydrate diet and 4 weeks traditional diet
  Difference of time spent in range (70-140 mg/dL) between the moderate carbohydrate diet and the traditional diet.
Time below range | 4 weeks moderate carbohydrate diet and 4 weeks traditional diet
  Difference of time spent below range (<70 mg/dL) between the moderate carbohydrate diet and the traditional diet.
Time in level 2 hypoglycemia | 4 weeks moderate carbohydrate diet and 4 weeks traditional diet
  Difference of time spent below range of 54 mg/dL between the moderate carbohydrate diet and the traditional diet.
Time above range | 4 weeks moderate carbohydrate diet and 4 weeks traditional diet
  Difference of time spent above range (>180 mg/dL) between the moderate carbohydrate diet and the traditional diet.
Time in level 2 hyperglycemia | 4 weeks moderate carbohydrate diet and 4 weeks traditional diet
  Difference of time spent above range of 250 mg/dL between the moderate carbohydrate diet and the traditional diet.
Hemoglobin A1c | 4 weeks moderate carbohydrate diet and 4 weeks traditional diet
  Difference of hemoglobin A1c between the moderate carbohydrate diet and the traditional diet.
Mean blood glucose | 4 weeks moderate carbohydrate diet and 4 weeks traditional diet
  Difference of mean blood glucose between the moderate carbohydrate diet and the traditional diet.
Glycemic variability: standard deviation and coefficient of variation | 4 weeks moderate carbohydrate diet and 4 weeks traditional diet
  Difference of glycemic variability, in terms of standard deviation (SD) and coefficient of variation (CV) of blood glucose levels between the moderate carbohydrate diet and the traditional diet.
Daily insulin dose | 4 weeks moderate carbohydrate diet and 4 weeks traditional diet
  Difference of insulin doses (total, basal and bolus) between the moderate carbohydrate diet and the traditional diet.
Number of severe hypoglycemic events | 4 weeks moderate carbohydrate diet and 4 weeks traditional diet
  Difference in the frequency of severe hypoglycemic events between the moderate carbohydrate diet and the traditional diet.
Number of diabetic ketoacidosis | 4 weeks moderate carbohydrate diet and 4 weeks traditional diet
  Difference in the frequence of diabetic ketoacidosis between the moderate carbohydrate diet and the traditional diet.
Body weight | 4 weeks moderate carbohydrate diet and 4 weeks traditional diet
  Difference in body weight between the moderate carbohydrate diet and the traditional diet.
Body mass index | 4 weeks moderate carbohydrate diet and 4 weeks traditional diet
  Difference in body mass index between the moderate carbohydrate diet and the traditional diet.
Blood lipids (total cholesterol, triglycerides, high density lipoprotein and low density lipoprotein concentrations) | 4 weeks moderate carbohydrate diet and 4 weeks traditional diet
  Difference in blood lipids (total cholesterol, triglycerides, high density lipoprotein and low density lipoprotein concentrations) between the moderate carbohydrate diet and the traditional diet.
Satisfaction with the diet in the context of diabetes treatment | 4 weeks moderate carbohydrate diet and 4 weeks traditional diet
  Difference in the satisfaction with the diet (Diabetes treatment satisfaction questionnaire - DTSQs) between the moderate carbohydrate diet and the traditional diet. The DTSQs has a scale of 0-48 and a higher score is associated with a higher treatment satifaction.
Bioelectrical impedance analysis | 4 weeks moderate carbohydrate diet and 4 weeks traditional diet
  Difference in bioelectrical impedance analysis between the moderate carbohydrate diet and the traditional diet.
Carb ratio | 4 weeks moderate carbohydrate diet and 4 weeks traditional diet
  Difference in carb ratio between the moderate carbohydrate diet and the traditional diet.
Active insulin time | 4 weeks moderate carbohydrate diet and 4 weeks traditional diet
  Difference in active insulin time between the moderate carbohydrate diet and the traditional diet.
Number of people who use glucose target 100 mg/dL, 110 mg/dL and 120 mg/dL | 4 weeks moderate carbohydrate diet and 4 weeks traditional diet
  Difference in umber of people who use glucose target 100 mg/dL, 110 mg/dL and 120 mg/dL between the moderate carbohydrate diet and the traditional diet.
Consumed carbohydrates | 4 weeks moderate carbohydrate diet and 4 weeks traditional diet
  Difference in consumed carbohydrates between the moderate carbohydrate diet and the traditional diet.
Meal composition | 4 weeks moderate carbohydrate diet and 4 weeks traditional diet
  Difference in meal composition a between the moderate carbohydrate diet and the traditional diet.

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Casteels, Prof, Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Vlaams-Brabant, Belgium